CLINICAL TRIAL: NCT03900143
Title: Safety, Efficacy and Usage Compliance of the Silk'n Tightra Home Use Device for Improvement of Sexual Functioning, Vulvovaginal Appearance and Reduction of SUI.
Brief Title: Safety, Efficacy and Usage Compliance of the Silk'n Tightra Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Home Skinovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO114314A
Record Dates: First submitted 2019-03-25; First posted 2019-04-02 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-03

CONDITIONS: Stress Urinary Incontinence; Sexual Dysfunction; Vulvovaginal Atrophy
MeSH Terms: conditions — Urinary Incontinence, Stress; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment - Tightra (Experimental): Treatment group with the Tightra device
  Interventions: Device: Tightra vaginal device

INTERVENTIONS:
Device: Tightra vaginal device — Vaginal device for improvement of vaginal symptoms, reduce vaginal laxity, improve sexual functioning, and treat stress urinary incontinence.

SUMMARY:
This is an open label, prospective study aimed to evaluate safety and efficacy of the Silk'n Tightra device for improvement of sexual functioning, vulvovaginal appearance and reduction of SUI.

DETAILED DESCRIPTION:
This is an open label, prospective study aimed to evaluate safety and efficacy of the Silk'n Tightra device.

The study includes 12 treatment sessions 3 times a week, over a period of 4 weeks. Each subject will serve as her own control, while comparing results before and after treatment. Treatment will be performed on the internal volva for 20 min according to the device instructions, .

Subjects that are interested in improving their labial appearance, and are willing to perform the external treatment twice a week in addition to the internal treatments, will be offered to conduct both treatments. The study will include one follow-up visit conducted one month following treatment end. During the second month of the study subjects will perform mainte-nance treatments and will gradually reduce the frequency of the treat-ments as follows:

* Week 5: 2 treatments
* Weeks 6-8: 1 treatment per week.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25-65 (at least 18 women in the range of 40-65 and approxi-mately 10 women in the range of 25 - 40)
2. The subject has symptoms of vaginal relaxation syndrome and uri-nary incontinence, and desires vaginal rejuvenation treatment.
3. The subject has had at least one vaginal delivery
4. The subject is sexually active.
5. The subject suffers from bad sexual functioning due to vaginal laxity and/or other vaginal symptoms.
6. Negative PAP smear and pelvic exam done within last 2 years.
7. The subjects should understand the information provided about the investigative nature of the treatment, possible benefits and side ef-fects, and sign the Informed Consent Form.
8. The subjects should be willing to comply with the study procedure and schedule, including the follow up visits.
9. The subject is able to read the User Manual.
10. Negative results in a urine pregnancy test

Exclusion Criteria:

1. Active electrical implant/device in any region of the body - Pacemak-er or internal defibrillator.
2. Presence of vulvar lesions or disease (dermatitis, human papilloma-virus, herpes simplex, vulvar dystrophy, etc.).
3. Superficial metal, piercing or other implants in the treatment area.
4. Vaginal or pelvic surgery or anti-incontinence surgery within the past 12 months.
5. Current urinary tract infection, pelvic or pelvic tract infection
6. Current cancer condition or pre-malignant moles.
7. History of skin and genital areas cancer.
8. Severe concurrent conditions, such as cardiac disorders, sensory dis-turbances, epilepsy, uncontrolled hypertension, and liver or kidney diseases, per investigator's discretion.
9. Pregnancy, nursing, or planned pregnancy within the next two months.
10. Prior labiaplasty
11. presence of major psychiatric conditions or related need for medica-tion
12. Diffuse pain syndrome or chronic pain requiring daily narcotics
13. Chronic use of anti-inflammatory agents (including steroids) and im-munosuppressants.
14. Undiagnosed abnormal genital bleeding
15. Presence of any condition or use of medication known to interfere with sexual activity
16. Poorly controlled endocrine disorders, such as Diabetes, or thyroid dysfunction and hormonal virilisation.
17. Isotretinoin (Accutane) within last 6 months.
18. Uterine prolapse, cystocele or rectocele.
19. History of bleeding coagulopathies, or use of anticoagulants except for low-dose aspirin.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only women should participate in this study
Enrollment: 28 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
An improvement in stress urinary incontinence | 8 weeks
  Improvement in SUI according to a validated questionnaire (ICIQ)
An improvement in stress urinary incontinence | 8 weeks
  Improvement in SUI according to a validated questionnaire (IIQ-7)

SECONDARY OUTCOMES:
improvement in sexual functioning | 8 weeks
  according to a validated questionnaire (FSFI)
Improvement in vaginal tightening (reduced laxity) and improvement in volvovaginal symptoms | 8 weeks
  According to a validated questionnaire.
Improvement in general satisfaction from the devcie | 8 weeks
  According to a satisfaction questionnaire
level of reduction in sexual distress | 8 weeks
  According to a validated questionnaire (FSDS)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Brandt, PhD, Principal Investigator — proDERM research institute
Locations (1):
- ProDERM, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No